CLINICAL TRIAL: NCT04524390
Title: Randomized, Double-Blind, Placebo-Controlled Phase 2 Study to Evaluate the Efficacy and Safety of Maralixibat in the Treatment of Subjects With Biliary Atresia After Hepatoportoenterostomy
Brief Title: Evaluation of Maralixibat in Biliary Atresia Response Post-Kasai
Acronym: EMBARK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRX-701
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Biliary Atresia
Keywords: Biliary Atresia; Kasai; Biliary Tract Diseases; Bile Duct Diseases; Congenital Abnormalities
MeSH Terms: conditions — Biliary Atresia; Biliary Tract Diseases; Bile Duct Diseases; Congenital Abnormalities | interventions — maralixibat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double Blind - Maralixibat (Experimental): The double-blind period comprised of 4-8 weeks of dose escalation followed by 18 - 22 weeks of stable dosing treatment, after which participants were transferred to the open-label arm.
  Interventions: Drug: Maralixibat
- Double Blind - Placebo (Placebo Comparator): The double-blind period comprised of 4-8 weeks of dose escalation followed by 18 - 22 weeks of stable dosing treatment, after which participants were transferred to the open-label arm.
  Interventions: Other: Placebo
- Open Label - Maralixibat (Experimental): The Open-Label period comprised of 4-8 weeks of dose escalation followed by 70 - 74 weeks of stable dosing treatment. During the OLE, all participants, regardless of treatment assignment in the double-blind period, received maralixibat.
  Interventions: Drug: Maralixibat

INTERVENTIONS:
Drug: Maralixibat — A small molecule inhibitor of the ileal bile acid transporter (IBAT)
  Other Names: Formerly LUM001 and SHP625
  Arms: Double Blind - Maralixibat; Open Label - Maralixibat
Other: Placebo — Identical to maralixibat except for the active drug substance
  Arms: Double Blind - Placebo

SUMMARY:
A study to evaluate the efficacy and safety of maralixibat in infants with Biliary Atresia (BA) after Hepatoportoenterostomy (HPE, also known as the Kasai procedure).

DETAILED DESCRIPTION:
This is a double-blind randomized, placebo-controlled study in subjects with Biliary Atresia with a primary endpoint at Week 26 followed by long-term open-label period during which all subjects will receive maralixibat to Week 104.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with body weight ≥2500 g, who are ≥21 days old and <90 days old at the time of HPE (Kasai)
2. HPE or Kasai Procedure within 3 weeks prior to randomization
3. Clinical diagnosis of biliary atresia

Exclusion Criteria:

1. Subjects with intractable chronic diarrhea at randomization
2. Subjects not tolerating enteral feeds at randomization
3. History of ileal resection
4. Diagnosis of biliary atresia splenic malformation syndrome or cystic biliary atresia
5. Evidence of another non-biliary atresia pathology involving the intrahepatic bile duct (e.g., paucity, sclerosing cholangitis)
6. Evidence of liver failure (e.g. significant ascites)

Ages: 21 Days to 111 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (7):
  - Phoenix Children's Division of Gastroenterology & Hepatology, Phoenix, Arizona
  - Children's Healthcare of Atlanta - Emory University School of Medicine, Atlanta, Georgia
  - NYU Grossman School of Medicine, New York, New York
  - New York-Presbyterian - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
- China (5):
  - Beijing Pediatric Research Institute, Beijing, Beijing Municipality
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - The Children's Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang
  - Children's hospital of Shanghai, Shanghai
  - Children's Hospital of Fudan University, Shanghai
- Hannover Medical School, Hanover, Germany
- Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw, Poland
- KK women's and Children's hospital, Bukit Timah, Singapore
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - King's College Hospital NHS, London
- Vietnam (3):
  - Hue Central Hospital, Huế, Thừa Thiên Huế Province
  - Vietnam National Children's Hospital, Hanoi
  - Children's Hospital No. 1, Ho Chi Minh City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 75 participants were enrolled at 19 sites across 8 countries (China, Germany, Poland, Singapore, Taiwan, United Kingdom, United States, and Vietnam).
Pre-assignment Details: The screening period starts when informed consent (by the legally authorized representative) is signed. The duration of the screening period is up to 3 weeks, during which all procedures listed for the screening visit in the schedule of assessment must be completed. A total of 77 patients were screened.
Period: Double Blind
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo | Open Label - Maralixibat
Started | 40 | 35 | 0
Completed | 28 | 24 | 0
Not Completed | 12 | 11 | 0
Not completed — Consent Withdrawal by subject | 2 | 1 | 0
Not completed — Adverse Event | 5 | 3 | 0
Not completed — Liver Transplant | 5 | 6 | 0
Not completed — Disease Progression | 0 | 1 | 0
Period: Open-Label
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo | Open Label - Maralixibat
Started | 0 | 0 | 52
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 51
Not completed — Drug interruption criteria | 0 | 0 | 1
Not completed — Liver Transplant | 0 | 0 | 1
Not completed — Disease Progression | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Study Termination by sponsor | 0 | 0 | 45

BASELINE CHARACTERISTICS:
Groups:
- Double Blind Period - Placebo; Double Blind - Maralixibat: The double-blind period comprised of 4-8 weeks of dose escalation followed by 18 - 22 weeks of stable dosing treatment.
- Total: Total of all reporting groups
Arm/Group | Double Blind Period - Placebo | Double Blind - Maralixibat | Total
Number analyzed (Participants) | 35 | 40 | 75
Age, Customized [Number; unit: participants]
  Infants and toddlers (28 days-23 months) | 35 | 40 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 20 | 19 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 28 | 31 | 59
  Race: White | 5 | 8 | 13
  Race: More than one race | 0 | 1 | 1
  Race: Not Reported | 1 | 0 | 1
  Race: Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Vietnam | 8 | 9 | 17
  Singapore | 0 | 1 | 1
  United States | 1 | 4 | 5
  China | 18 | 18 | 36
  Taiwan | 1 | 2 | 3
  Poland | 1 | 1 | 2
  United Kingdom | 6 | 4 | 10
  Germany | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Total Serum Bilirubin Levels
Time Frame: From baseline to Week 26
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo
Number analyzed (Participants) | 40 | 35
mg/dl | -3.5 (0.853) | -3.11 (0.947)
Statistical Analysis 1: Comparison: Double Blind - Maralixibat vs Double Blind - Placebo; Test type: Superiority; p = 0.7419, MMRM; Least-Square mean = -0.39, 95% CI 2-sided [-2.76 to 1.97], Standard Error of Mean 1.182

2. Secondary Outcome: Mean Change in Total Serum Bile Acids
Time Frame: From baseline to Week 26
Measure: Least Squares Mean (Standard Error); unit: umol/L
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo
Number analyzed (Participants) | 40 | 35
umol/L | -51.19 (24.436) | -5.29 (28.440)
Statistical Analysis 1: Comparison: Double Blind - Maralixibat vs Double Blind - Placebo; Test type: Superiority; p = 0.2002, MMRM; Least-Square mean = -45.9, 95% CI 2-sided [-116.86 to 25.05], Standard Error of Mean 35.398

3. Secondary Outcome: Proportion of Participants With Mean TSB Levels <2 mg/dL Through Week 26
Time Frame: From baseline to Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo
Number analyzed (Participants) | 40 | 35
Participants | 24 | 20
Statistical Analysis 1: Comparison: Double Blind - Maralixibat vs Double Blind - Placebo; Test type: Superiority; p = 0.8412, Barnard's exact test

4. Secondary Outcome: Proportion of Participants Observed to Have a Liver-related Clinical Event Transplantation, Liver Decompensation, Discontinuations Due to Liver Related Events, or Death.
Description: Liver decompensation (hepatic encephalopathy, variceal bleeding, new persistent ascites)
Time Frame: From Baseline to Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo
Number analyzed (Participants) | 40 | 35
Participants | 8 | 7
Statistical Analysis 1: Comparison: Double Blind - Maralixibat vs Double Blind - Placebo; Test type: Superiority; p > 0.9999, Barnard's exact test

5. Secondary Outcome: Proportion of Participants Undergoing Liver Transplantation or Death
Time Frame: From Baseline to Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo
Number analyzed (Participants) | 40 | 35
Participants | 5 | 3
Statistical Analysis 1: Comparison: Double Blind - Maralixibat vs Double Blind - Placebo; Test type: Superiority; p = 0.6658, Barnard's exact test

6. Secondary Outcome: Proportion of Participants Observed to Develop Clinically Evident Portal Hypertension Defined as Splenomegaly and Thrombocytopenia (Platelet Count <150 x 109/L) or Clinically Evident Ascites or Endoscopic Evidence of Esophageal or Gastric Varices.
Description: Splenomegaly => (spleen size >2 cm below the costal margin palpated on physical examination)
Time Frame: From Baseline to Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo
Number analyzed (Participants) | 40 | 35
Participants | 3 | 4
Statistical Analysis 1: Comparison: Double Blind - Maralixibat vs Double Blind - Placebo; Test type: Superiority; p = 0.6236, Barnard's exact test

7. Secondary Outcome: Proportion of Participants With Mean TSB Levels ≤1.2 mg/dL
Time Frame: From Baseline to Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo
Number analyzed (Participants) | 40 | 35
Participants | 23 | 18
Statistical Analysis 1: Comparison: Double Blind - Maralixibat vs Double Blind - Placebo; Test type: Superiority; p = 0.6658, Barnard's exact test

8. Secondary Outcome: Proportion of Participants With Mean sBA Levels ≤40 mmol/L
Time Frame: From Baseline to Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo
Number analyzed (Participants) | 40 | 35
Participants | 10 | 7
Statistical Analysis 1: Comparison: Double Blind - Maralixibat vs Double Blind - Placebo; Test type: Superiority; p = 0.6659, Barnard's exact test

ADVERSE EVENTS:
Time Frame: Baseline to EOT. In this study the longest time frame was 102.4 weeks
Groups:
- Double Blind - Maralixibat: All participants who receive at least 1 dose of study medication during the double-blinded Maralixibat Period.
- Double Blind - Placebo: All participants who receive at least 1 dose of study medication during the double-blinded Placebo Period.
- Open Label - Maralixibat: All participants who receive at least 1 dose of study medication during the Open-Label Maralixibat Period.
Arm/Group | Double Blind - Maralixibat | Double Blind - Placebo | Open Label - Maralixibat
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/35 | 0/52
Serious Adverse Events (participants affected / at risk) | 26/40 | 25/35 | 21/52
Other Adverse Events (participants affected / at risk) | 38/40 | 33/35 | 47/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind - Maralixibat (N=40) | Double Blind - Placebo (N=35) | Open Label - Maralixibat (N=52)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 15 (23) | 17 (25) | 8 (10)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (13) | 4 (5) | 2 (2)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hyperinsulinism (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind - Maralixibat (N=40) | Double Blind - Placebo (N=35) | Open Label - Maralixibat (N=52)
Alanine aminotransferase increased (Investigations) | 5 (5) | 5 (5) | 4 (6)
Blood bilirubin increased (Investigations) | 1 (3) | 2 (2) | 1 (1)
Hepatic enzyme increased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Spleen palpable (Investigations) | 0 (0) | 2 (2) | 1 (1)
Vitamin A decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (5) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 2 (3) | 3 (4) | 2 (3)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 14 (19) | 8 (8) | 12 (18)
Diarrhoea (Gastrointestinal disorders) | 13 (19) | 8 (8) | 13 (16)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (8) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 6 (8) | 6 (6) | 3 (3)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (6) | 8 (9)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (6) | 0 (0) | 5 (8)
Eczema (Skin and subcutaneous tissue disorders) | 6 (9) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 3 (3) | 4 (5)
COVID-19 (Infections and infestations) | 3 (3) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (7)
Otitis media (Infections and infestations) | 0 (0) | 1 (2) | 3 (3)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 6 (8) | 5 (8) | 5 (6)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 3 (5) | 12 (23)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (5) | 4 (6)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Parainfluenzae virus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Vitamin A deficiency (Metabolism and nutrition disorders) | 3 (3) | 7 (7) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 (7) | 9 (9) | 8 (8)
Vitamin E deficiency (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 4 (4)
Zinc deficiency (Metabolism and nutrition disorders) | 5 (5) | 5 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT04524390/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT04524390/SAP_001.pdf